CLINICAL TRIAL: NCT03709316
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Phase III Clinical Trial Evaluating the Efficacy and Safety of ZL-2306 (Niraparib) for Maintenance Treatment in Patients With Advanced Ovarian Cancer, Fallopian Tube Carcinoma or Primary Peritoneal Cancer (Collectively Referred to as Ovarian Cancer) Who Have Achieved Effective Response After First-line Platinum-containing Chemotherapy
Brief Title: A Study of ZL-2306 (Niraparib) as Maintenance Treatment Following First-line Chemotherapy in Patients With Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZL-2306-004
Record Dates: First submitted 2018-09-19; First posted 2018-10-17 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZL-2306 (Nirapairb) (Experimental): The starting dose is 300mg or 200mg QD based on the subject's baseline body weight or baseline platelet count
  Interventions: Drug: ZL-2306 (Nirapairb)
- Placebo (Placebo Comparator): The starting dose is 300mg or 200mg QD based on the subject's baseline body weight or baseline platelet count
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: ZL-2306 (Nirapairb) — The starting dose is 300mg or 200mg QD based on the subject's baseline body weight or baseline platelet count
  Arms: ZL-2306 (Nirapairb)
Drug: Placebo Comparator — The starting dose is 300mg or 200mg QD based on the subject's baseline body weight or baseline platelet count
  Arms: Placebo

SUMMARY:
Niraparib is a PARP inhibitor. This is a 2:1 randomized, double-blind, placebo-controlled study conducted in patients with advanced (FIGO Stage III or IV) ovarian cancer to evaluate Efficacy and Safety of ZL-2306 (Niraparib) for Maintenance Treatment

ELIGIBILITY:
Inclusion Criteria:

* 1. The written informed consent form shall be signed before proceeding with any study-related procedure.
* 2. The subject agrees to collection of blood samples for detection of gBRCA mutations (gBRCA mutation status must be known before randomization).
* 3. The subject shall be a female, aged 18 years or older.
* 4. Histologically confirmed high-grade serous/endometrioid or dominantly high-grade serous/endometrioid epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinoma (no histological restriction for patients carrying germline BRCA mutations).

Note: Patients who have received neoadjuvant chemotherapy can also be enrolled if their tumors after chemotherapy cannot be pathologically graded.

* 5. FIGO staging is Stage III or IV.
* 6. Criteria for previous surgery (meeting any of these):

  * Inoperable Stage III or IV patients
  * Stage IV patients, regardless of postoperative residual lesion status
  * Stage III patients who have undergone primary tumor reductive surgery with postoperative residual lesion status of R1 (microscopic residual lesions) or R2 (macroscopic residual lesions)
  * Stage III or IV patients who have undergone intermittent tumor reductive surgery (patients who have used neoadjuvant therapy) regardless of postoperative residual lesion status
* 7. Criteria for previous chemotherapy:

  * It is allowed to enroll patients who have received intraperitoneal chemotherapy
  * Patients have completed at least 6 cycles yet no more than 9 cycles of first-line platinum-containing chemotherapy (preferably carboplatin, but cisplatin is also acceptable)
  * Patients undergoing intermittent tumor reductive surgery should respectively receive at least 2 cycles of platinum-containing chemotherapy preoperatively and postoperatively, and receive a total of at least 6 cycles yet no more than 9 cycles of chemotherapy (preferably carboplatin, but cisplatin is also acceptable) preoperatively and postoperatively
  * Patients are assessed by the investigator to have achieved complete response (CR) or partial response (PR) after first-line platinum-containing chemotherapy, and the efficacy assessment should be performed after the end of at least 3 cycles of chemotherapy
  * CA-125 level must be within the normal range after the end of chemotherapy or has decreased by more than 90% during the course of first-line chemotherapy and remains so for at least 7 days (the elevation of CA-125 prior to enrollment shall not exceed 15% compared with the CA-125 level after the end of chemotherapy)
  * Patients must be randomized within 12 weeks since Day 1 of the last cycle of chemotherapy 8. Patients must be able to submit formalin-fixed, paraffin-embedded tumor tissue samples.
* 9. ECOG physical condition score of the patient shall be 0 or 1.
* 10. Organ function is in good condition, including:

  * Neutrophil count ≥1.5×109/L
  * Platelet count ≥100×109/L
  * Hemoglobin ≥100 g/L
  * Serum creatinine is not more than 1.5 times the normal upper limit, or creatinine clearance rate is not less than 60 mL/min (calculated with Cockcroft-Gault formula)
  * Total bilirubin is not more than 1.5 times the normal upper limit, or direct bilirubin is not more than 1.0 time the normal upper limit.
  * AST and ALT are not more than 2.5 times their normal upper limit, and with existence of hepatic metastasis, these values must not be more than 5 times their normal upper limit.
* 11. Only the female patient who has been tested with pregnancy-negative result and had made a commitment to adopt effective contraption measures or to avoid sexual behavior from the start to the completion of the study and within 3 months after the last administration of study medication is eligible to be enrolled into the study. Or female patients without childbearing potential may be enrolled in the study, defined as follows:

  * A female who has undergone surgical birth control operation (e.g., hysterectomy, bilateral ovariectomy, or bilateral tubal resection); or
  * A female aged 60 years or older; or
  * A female, aged ≥40 years and <60 years, with a period of menolipsis for 12 months or longer, whose follicle-stimulating hormone test results are within the post-menopause reference range of the study institution.
* 12. Patients must be able to take medication orally and have the ability to comply with the protocol.
* 13. Any previous toxic and side effect of the patient has restored to CTCAE grade ≤1 or the baseline level, except for CTCAE grade ≤2 symptomatically stable sensory neuropathy or alopecia.

Exclusion Criteria:

* 1. Patients diagnosed with mucinous, clear cell subtypes of epithelial ovarian cancer, carcinosarcoma, or undifferentiated ovarian cancer.
* 2. Stage III patients who have undergone primary tumor reductive surgery with postoperative status of R0-complete resection (with no residual lesion).
* 3. Patients who have undergone tumor reductive surgery more than twice.
* 4. Patients who plan to or have used bevacizumab as maintenance therapy after first-line platinum-containing chemotherapy. If the patient received bevacizumab in platinum-containing chemotherapy but did not receive bevacizumab as maintenance therapy, and the last dose of bevacizumab was used ≥ 28 days before signing the master informed consent form, the patient can be enrolled.
* 5. Patients who are known to be allergic to active or inactive ingredients of ZL-2306 (niraparib) or other drugs with similar chemical structures to ZL-2306 (niraparib).
* 6. Patients who have previously been treated with PARP inhibitors (including niraparib).
* 7. Patients who have received other study drug treatment within 4 weeks prior to the first administration or < 5 elimination half-lives of the study drug (whichever is longer).
* 8. Patients with ≥ grade 3 anemia, neutropenia or thrombocytopenia due to prior chemotherapy for more than 4 weeks.
* 9. Patients with transfusion-dependent anemia or thrombocytopenia, including:

  * Patients who have received blood transfusion (platelet or red blood cell) within 2 weeks before the first dose
  * Patients who have received colony stimulating factor therapy (e.g., granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF), or recombinant erythropoietin) within 2 weeks before the first dose
* 10. Patients who have undergone ascites drainage within 4 weeks prior to enrollment.
* 11. Brain metastases or leptomeningeal metastases that have not been treated or whose symptoms have not been controlled (e.g., new or worsening symptoms or signs, or the required dose of hormones is not yet stable). Note: It is not necessary to perform an imaging scan to confirm whether there is a brain metastasis or not; patients with spinal cord compression who have received symptomatic treatment and have evidence on clinical stable status of the disease for at least 28 days could still be considered as eligible for enrollment.
* 12. Patients who have received a major surgery 3 weeks before the start of the study, or is subject to any surgical effect that has not yet been recovered after surgery.
* 13. Patients who have received palliative radiotherapy for > 20% of bone marrow 3 weeks prior to enrollment.
* 14. Patients suffered from invasive cancers other than ovarian cancer within 5 years prior to enrollment (except for treated carcinoma in situ of cervix, non-melanoma and ductal carcinoma in situ).
* 15. Patients who have been diagnosed previously or currently with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* 16. Patients who have got other severe or uncontrollable diseases, including but not limited to:

  * Hardly controllable nausea and vomiting, inability to swallow the study drug, and any gastrointestinal disease that may interfere with the absorption and metabolism of the drug
  * Human immunodeficiency virus (HIV) infection, active hepatitis (hepatitis B, hepatitis C)
  * Uncontrolled ventricular arrhythmias, myocardial infarction that occurred within 3 months before enrollment
  * Uncontrollable grand mal epilepsy, unstable spinal cord compression, superior vena cava syndrome or other psychiatric disorders that may affect signing of the informed consent by the patient
  * Immunodeficiency (except for splenectomy), or other diseases which, as believed by investigators, could expose the patient to a high risk
* 17. Patients who are pregnant or breastfeeding currently, or expect to plan for pregnancy in the course of the study treatment.
* 18. The corrected QT interval (QTc) is more than 470 msec; if the patient has an extended QTc interval, but investigators find such a extension is caused by a cardiac pacemaker (without any other cardiac abnormality), it shall be necessary to determine whether the patient is eligible for enrollment or not based on the discussion with the study physician from the sponsor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 384 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2022-01-29 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
BICR-assessed progression-free survival (PFS) | Approximately 36 months since the first subject enrolled
  the time from randomization to progressive disease or death due to various causes assessed by the BICR according to RECIST 1.1, whichever occurs first

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 36 months since the first subject enrolled
  the time from the date of randomization to the date of death caused by any reason.
Time to first subsequent anti-tumor treatment (TFST) | Approximately 36 months since the first subject enrolled
  the time from the date of randomization in the study to the date when the first subsequent anti-tumor treatment starts
PFS and OS assessed by BICR in patients with HRD (homologous recombination defects) | Approximately 36 months since the first subject enrolled
  positive patient population (including gBRCA-positive patients).

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Anhui Provincal Hospital, Hefei, Anhui
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The first affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guizhou Cancer hospital, Guiyang, Guizhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan hospital of wuhan university, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - second hospital of Shanxi medical university, Taiyuan, Shanxi
  - West China second university hospital, Chengdu, Sichuan
  - Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, Tianjin Municipality
  - Affiliate Cancer Hospital Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Woman's hospital School of medicine Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - the First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital of Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Tumour Hospital, Tianjin

REFERENCES:
- [Derived] Li N, Zhu J, Yin R, Wang J, Pan L, Kong B, Zheng H, Liu J, Wu X, Wang L, Huang Y, Wang K, Zou D, Zhao H, Wang C, Lu W, Lin A, Lou G, Li G, Qu P, Yang H, Zhang Y, Cai H, Pan Y, Hao M, Liu Z, Cui H, Yang Y, Yao S, Zhen X, Hang W, Hou J, Wang J, Wu L. Treatment With Niraparib Maintenance Therapy in Patients With Newly Diagnosed Advanced Ovarian Cancer: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2023 Sep 1;9(9):1230-1237. doi: 10.1001/jamaoncol.2023.2283. PMID 37440217